CLINICAL TRIAL: NCT06164717
Title: Behavioral and Neural Characteristics of Adaptive Speech Motor Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ludo Max, Professor, Department of Speech and Hearing Sciences, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001367; R01DC020707 (NIH); R01DC014510 (NIH)
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Speech
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auditory feedback perturbation during speech (Experimental): The intervention consists of manipulating real-time auditory feedback during speech production. In our lab, such feedback perturbations can be implemented with either a stand-alone digital vocal processor (a device commonly used by singers and the music industry) or with software-based signal processing routines (see Equipment section for details). Note that the study does not investigate the efficacy of these hardware or software methods to induce behavioral change in subjects' speech. Rather, the study addresses basic experimental questions regarding the general role of auditory feedback in the central nervous system's control of articulatory speech movements.
  Interventions: Behavioral: Auditory feedback perturbation during speech
- Visual feedback perturbation during reaching (Experimental): The intervention consists of manipulating real-time visual feedback during upper limb reaching movements. In our lab, such feedback perturbations can be implemented with a virtual reality display system.
  Interventions: Behavioral: Visual feedback perturbation during reaching
- Deep brain stimulation (Experimental): This intervention consists of toggling the deep brain stimulation (DBS) implant ON/OFF prior to participation in the speech auditory-motor learning tasks and speech sequence learning tasks. This intervention can be implemented by the subject themselves as all patients have a hand- held controlled that they use to switch stimulation ON/OFF.
  Interventions: Other: DBS stimulation ON/OFF

INTERVENTIONS:
Behavioral: Auditory feedback perturbation during speech — The intervention consists of manipulating real-time auditory feedback during speech production. In our lab, such feedback perturbations can be implemented with either a stand-alone digital vocal processor (a device commonly used by singers and the music industry) or with software-based signal processing routines (see Equipment section for details). Note that the study does not investigate the efficacy of these hardware or software methods to induce behavioral change in subjects' speech. Rather, the study addresses basic experimental questions regarding the general role of auditory feedback in the central nervous system's control of articulatory speech movements.
  Arms: Auditory feedback perturbation during speech
Behavioral: Visual feedback perturbation during reaching — The intervention consists of manipulating real-time visual feedback during upper limb reaching movements. In our lab, such feedback perturbations can be implemented with a virtual reality display system.
  Arms: Visual feedback perturbation during reaching
Other: DBS stimulation ON/OFF — Patients who have been previously implanted with a DBS stimulator for their clinical care will be tested in two speech motor learning tasks with the stimulation ON and with the stimulation OFF.
  Note that (1) patients routinely turn the stimulation OFF and back ON (examples are, for some patients, to sleep, to save battery, etc), and (2) we are not in any way evaluating the stimulator itself or its clinical effectiveness but only whether or not two forms of speech motor learning (adaptation to auditory feedback perturbation and speech sequence learning) are affected differently by having the stimulation ON or OFF.
  implant ON/OFF prior to participation in the speech auditory-motor learning tasks and speech sequence learning tasks. This intervention can be implemented by the subject themselves as all patients have a hand- held controlled that they use to switch stimulation ON/OFF.
  Arms: Deep brain stimulation

SUMMARY:
This study meets the NIH definition of a clinical trial, but is not a treatment study. Instead, the goal of this study is to investigate how hearing ourselves speak affects the planning and execution of speech movements. The study investigates this topic in both typical speakers and in patients with Deep Brain Stimulation (DBS) implants. The main questions it aims to answer are:

* Does the way we hear our own speech while talking affect future speech movements?
* Can the speech of DBS patients reveal which brain areas are involved in adjusting speech movements? Participants will read words, sentences, or series of random syllables from a computer monitor while their speech is being recorded. For some participants, an electrode cap is also used to record brain activity during these tasks. And for DBS patients, the tasks will be performed with the stimulator ON and with the stimulator OFF.

ELIGIBILITY:
General inclusion criteria:

* native speaker of American English
* no communication or neurological problems (except for subjects in the DBS group)
* 250-4000 Hz pure tone hearing thresholds equal to or better than 25 dB HL for children and young adults and equal to or better than 35 dB HL for older adults
* no medications that affect sensorimotor functioning (except for in the DBS group)
* adult subjects: 18 years of age or older
* typical children: 4;0 to 6;11 [years;months] or 10;0 to 12;11 [years;months])

Specific inclusion criteria for children:

* scoring above the 20th percentile on the Peabody Picture Vocabulary Test (PPVT-5), Expressive Vocabulary Test (EVT-3), Goldman-Fristoe Test of Articulation (GFTA-3), and either Test of Early Language Development (TELD-4) or (for children age 8 or older) Clinical Evaluation of Language Fundamentals (CELF-5).

Specific inclusion criteria for DBS patients:

* bilateral electrodes implanted in either the ventral intermediate nucleus of the thalamus (Vim; a target site for patients with essential tremor) or subthalamic nucleus (STN; a target site for patients with Parkinson's disease)

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 507 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Speech formant frequencies | Measurements will be made only from acoustic recordings made during the test session (~1 hour).
  The frequencies of the subject's first two formants (F1, F2) for each test word will be measured from spectrographic displays with overlaid Linear Predictive Coding formant tracks.
Reach direction for arm movements | Outcome measures will be made only during a single data recording session (~2 hours).
  Measuring initial reach direction for arm movements allows us to measure the direction that was planned before movement onset.
Amplitude of long-latency auditory evoked potentials (from EEG recordings) responses | Measurements will be made only from electroencephalography (EEG) recordings made during the test session (~2 hours).
  Amplitude of the N1 component (in microvolt) will be measured in response to both probe tones and to a subject's own speech onset.
Local field potentials recorded by neural implants | Measurements will be made only from DBS implant recordings made during the test session (~1-2 hours).
  Local field potentials (LFPs) will be recorded by the PerceptPC DBS implants and used to measure changes in power spectrum density across different phases of the tasks. Additionally, LFPs will be used to conduct event-related analyses.
Temporal measures of speech syllable sequence learning | Outcome measures will be made only during a single data recording session (~0.5 hours)
  1. Speech onset time (in milliseconds); 2. Average syllable duration (in milliseconds)
Accuracy during speech syllable sequence learning | Outcome measures will be made only during a single data recording session (~0.5 hours)
  Sequence accuracy (in percent)

CONTACTS AND LOCATIONS:
Overall Officials: Ludo Max, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States